CLINICAL TRIAL: NCT05623020
Title: AN OPEN-LABEL, 2-ARM, MULTICENTER, RANDOMIZED PHASE 3 STUDY TO EVALUATE THE EFFICACY AND SAFETY OF ELRANATAMAB (PF-06863135) + DARATUMUMAB + LENALIDOMIDE VERSUS DARATUMUMAB + LENALIDOMIDE + DEXAMETHASONE IN TRANSPLANT-INELIGIBLE OR TRANSPLANT-DEFERRED PARTICIPANTS WITH NEWLY DIAGNOSED MULTIPLE MYELOMA
Brief Title: A Study to Learn About Effects of the Combination of Elranatamab, Daratumumab and Lenalidomide Compared With Daratumumab, Lenalidomide, and Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma Who Are Not Candidates for Transplant or Who Will Not Receive a Transplant as Initial Therapy
Acronym: MagnetisMM-6
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1071006; MAGNETISMM-6 (Other: Alias Study Number); 2024-514139-50-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-10-26; First posted 2022-11-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Elranatamab; PF-06863135; B-Cell Maturation Antigen; Daratumumab; Lenalidomide; Multiple myeloma; MagnetisMM-6
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Part 1, Dose Level 1: Elranatamab + Daratumumab + Lenalidomide (Experimental)
  Interventions: Drug: Elranatamab; Drug: Daratumumab; Drug: Lenalidomide
- Part 1, Multiple Dose Levels, Elranatamab + Daratumumab + Lenalidomide (Experimental)
  Interventions: Drug: Elranatamab; Drug: Daratumumab; Drug: Lenalidomide
- Part 2 Randomized Arm A: Elranatamab + Daratumumab + Lenalidomide (Experimental)
  Interventions: Drug: Elranatamab; Drug: Daratumumab; Drug: Lenalidomide
- Part 2 Randomized Arm B: Daratumumab + Lenalidomide + Dexamethasone (Active Comparator)
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone
- Part 1: Elranatamab + Lenalidomide (Experimental)
  Interventions: Drug: Elranatamab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Elranatamab — Part 1 Dose Level 1 is not randomized. All other cohorts are randomized.
  Arms: Part 1, Dose Level 1: Elranatamab + Daratumumab + Lenalidomide; Part 1, Multiple Dose Levels, Elranatamab + Daratumumab + Lenalidomide; Part 1: Elranatamab + Lenalidomide; Part 2 Randomized Arm A: Elranatamab + Daratumumab + Lenalidomide
Drug: Daratumumab — Part 1 Dose Level 1 is not randomized. All other cohorts are randomized.
  Arms: Part 1, Dose Level 1: Elranatamab + Daratumumab + Lenalidomide; Part 1, Multiple Dose Levels, Elranatamab + Daratumumab + Lenalidomide; Part 2 Randomized Arm A: Elranatamab + Daratumumab + Lenalidomide; Part 2 Randomized Arm B: Daratumumab + Lenalidomide + Dexamethasone
Drug: Lenalidomide — Part 1 Dose Level 1 is not randomized. All other cohorts are randomized.
Drug: Dexamethasone — Randomized
  Arms: Part 2 Randomized Arm B: Daratumumab + Lenalidomide + Dexamethasone

SUMMARY:
Elranatamab is a bispecific antibody: binding of elranatamab to CD3-expressing T-cells and BCMA-expressing multiple myeloma cells causes targeted T-cell-mediated cytotoxicity. The main purpose of the study is to evaluate if the combination of Elranatamab, Daratumumab and Lenalidomide offers superior clinical benefit compared with the combination of Daratumumab, Lenalidomide and Dexamethasone in people with newly diagnosed multiple myeloma.

There are 2 parts to this study. Part 1 will characterize the safety and tolerability of elranatamab in combination with daratumumab and lenalidomide or in combination with lenalidomide and will identify the optimal dose(s) of the combination regimen. Part 2 of the study will evaluate the minimal residual disease (MRD) negativity rate and the progression free survival (PFS) of the combination of elranatamab, daratumumab, and lenalidomide compared with the combination of daratumumab, lenalidomide, and dexamethasone in participants with newly diagnosed multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma (MM) as defined by IMWG criteria (Rajkumar et al., 2014)
* Measurable disease based on IMWG criteria as defined by at least 1 of the following:

  * Serum M-protein ≥0.5 g/dL;
  * Urinary M-protein excretion ≥200 mg/24 hours;
  * Involved FLC ≥10 mg/dL (≥100 mg/L) AND abnormal serum immunoglobulin kappa to lambda FLC ratio (<0.26 or >1.65).
* Part 1: Participants with relapsed/refractory multiple myeloma (RRMM) who have received 1-2 prior lines of therapy including at least one immunomodulatory drug and one proteasome inhibitor: or participants with newly-diagnosed multiple myeloma (NDMM) that are transplant-ineligible as defined by age ≥65 years or transplant-ineligible as defined by age <65 years with comorbidities impacting the possibility of transplant.
* Part 2: participants with newly-diagnosed multiple myeloma that are
* transplant-ineligible (defined by age or comorbidities impacting the possibility of transplant) or
* transplant deferred (defined as clinically transplant-eligible but who does not intend to receive transplant as a first line of therapy).
* ECOG performance status ≤2.
* Not pregnant and willing to use contraception
* For participants with RRMM: Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤1.

Exclusion Criteria:

* Smoldering Multiple Myeloma.
* Monoclonal gammopathy of undetermined significance.
* Waldenströms Macroglobulinemia
* Plasma cell leukemia.
* Active, uncontrolled bacterial, fungal, or viral infection, including (but not limited to) COVID-19/SARS-CoV-2, HBV, HCV, and known HIV or AIDS-related illness.
* Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ, or Stage 0/1 with minimal risk of recurrence per investigator.
* For participants with RRMM: Previous treatment with a BCMA-directed therapy or anti-CD38-directed therapy within 6 months preceding the first dose of study intervention in this study. Stem cell transplant ≤3 months prior to first dose of study intervention or active GVHD.
* For participants with NDMM: Previous systemic treatment for MM except for a short course of corticosteroids (ie, total of 160 mg dexamethasone or equivalent before the first dose of study intervention). A cumulative dose of systemic corticosteroids equivalent to ≥20 mg of dexamethasone during screening.
* Live attenuated vaccine administered within 4 weeks of the first dose of study intervention.
* Administration of investigational product (eg, drug or vaccine) concurrent with study intervention or within 30 days (or as determined by the local requirement) preceding the first dose of study intervention used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2030-10-18 (Estimated); Study Completion 2033-10-03 (Estimated)

PRIMARY OUTCOMES:
Part 1 Dose Limiting Toxicity | From the first dose of elranatamab/first full dose in combination with EDR until 28 days (+/- visit window) from the first administration of elranatamab with daratumumab and lenalidomide
Part 2: Progression free survival per IMWG | From randomization up to 97 months.
Part 2: Minimal Residual Disease negativity rate | At 12 months after randomization

SECONDARY OUTCOMES:
Overall Survival | From date of randomization up to 97 months
Overall minimal residual disease negativity rate | From date of randomization up to 97 months
Sustained MRD negativity rate (Part 2) | From date of randomization up to 97 months
Duration of minimal residual disease negativity (Part 2) | From date of minimal residual disease negative status up to 97 months
PFS by investigator | From date of randomization up to 97 months
PFS2 by investigator (Part 2) | From the date of randomization up to 97 months
Objective Response Rate | From the date of randomization up to 97 months
Complete Response Rate | From the date of randomization up to 97 months
Time to Response | From the date of randomization to date of confirmed objective response up to 97 months
Duration of Response | From the date of confirmed objective response up to 97 months
Duration of Complete Response | From the date of confirmed complete response up to 97 months
Frequency of treatment-emergent adverse events | From the date of first dose of study intervention up to 97 months
Frequency of abnormal laboratory results | From the date of first dose of study intervention up to 97 months
Pharmacokinetics of elranatamab when used in the elranatamab + daratumumab + lenalidomide or elranatamab + lenalidomide combinations | From date of first dose of study intervention up to 97 months
  Predose and post dose concentrations of elranatamab
Incidence of Anti-Drug Antibody against elranatamab | From date of first dose of study intervention up to 97 months
  Immunogenicity of elranatamab
Pharmacokinetics of daratumumab and lenalidomide when used in the elranatamab+daratumumab+lenalidomide or elranatamab+lenalidomide combinations (Part 1) | From date of first dose of study intervention up to 97 months
  Predose concentrations of daratumumab and lenalidomide
Health-related quality of life by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (Part 2) | From date the informed consent is signed up to 97 months
  Higher scores on the functional scales represent higher levels of functioning. Higher scores on the global health status/quality of life scale represent higher health status/quality of life. Higher scores on the symptom scales/items represent a greater presence of symptoms.
Health-related quality of life by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire -Myeloma 20 (Part 2) | From date the informed consent is signed up to 97 months
  Higher scores on the functioning subscales (body image, future perspective) represent higher levels of functioning, whereas higher scores on the symptom subscales (disease symptoms, side effects) represent a greater presence of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (85):
- Australia (4):
  - Pindara Private Hospital, Benowa, Queensland
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Epworth Freemasons, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Canada (3):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre, Toronto, Ontario
- China (11):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The first hospital of jilin university, Changchun, Jilin
  - Tongji University - Shanghai Fourth People's Hospital, Shanghai, Shanghai Municipality
  - Institute of hematology&blood disease hospital, Tianjin, Tianjin Municipality
  - The first Affiliated hospital of Wenzhou medical University, Wenzhou, Zhejiang
- Czechia (3):
  - Fakultní nemocnice Brno Bohunice, Brno, Brno-město
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (3):
  - Institut Universitaire du Cancer Toulouse - Oncopole - CHU de TOULOUSE, Toulouse, Haute-garonne
  - Centre Hospitalier Universitaire de Poitiers, Poitiers, Vienne
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes
- Germany (2):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Klinikum Chemnitz, Chemnitz
- Greece (4):
  - Evangelismos General Hospital of Athens, Athens, Attikí
  - Alexandra General Hospital of Athens, Athens, Attikí
  - "Theagenio" Cancer Hospital of Thessaloniki, Thessaloniki, Kentrikí Makedonía
  - University Hospital of Ioannina, Ioannina, Ípeiros
- Israel (5):
  - Rabin Medical Center, Petah Tikva, Central District
  - The Edmond and Lily Safra Children's HospitalnThe Chaim Sheba Medical CenternDepartment of Pediatric, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Soroka Medical Center, Beersheba, Southern District
  - Sourasky Medical Center, Tel Aviv, TELL ABĪB
- Italy (13):
  - AUSL di Piacenza, Piacenza, Emilia-Romagna
  - Ospedale Santa Maria delle Croci, Ravenna, Emilia-Romagna
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - Cro-Irccs, Aviano, Friuli Venezia Giulia
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardy
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Turin, Piedmont
  - A.O.U. Policlinico Paolo Giaccone, Palermo, Sicily
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Istituto Europeo di Oncologia IRCCS, Milan
  - ASL PESCARA-Presidio Ospedaliero Pescara, Pescara
  - Azienda Sanitaria Locale di Pescara, Pescara
  - AOU Policlinico Umberto I, Roma
- Japan (10):
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - Gunma University Hospital, Maebashi, Gunma
  - Iwate Medical University Hospital, Yahaba-cho, Iwate
  - Tohoku University Hospital, Sendai, Miyagi
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Yamagata University Hospital, Yamagata
- Albert Schweitzer Ziekenhuis, locatie Dordwijk, Dordrecht, South Holland, Netherlands
- Poland (3):
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw, Lower Silesian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Pratia Onkologia Katowice, Katowice, Silesian Voivodeship
- South Korea (7):
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [incheon]
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeonranamdo
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital(Seoul St. Mary's Hospital), Seoul, Seoul-teukbyeolsi [seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [seoul]
- Spain (11):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [LA Coruña]
  - Institut Català d'Oncologia (ICO) - Badalona, Badalona, Barcelona [barcelona]
  - Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet Del Llobregat, Barcelona [barcelona]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [cataluña]
  - Institut Català d'Oncologia (ICO) - Girona, Girona, Girona [gerona]
  - Clinica Universidad de Navarra, Madrid, Madrid, Comunidad de
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Doctor Peset, Valencia, València
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital La Princesa, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
- Kantonsspital Winterthur, Winterthur, Switzerland
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071006